CLINICAL TRIAL: NCT04435184
Title: Crizanlizumab for Treating COVID-19 Vasculopathy
Acronym: CRITICAL
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: Novartis (Industry); Socar Research SA (Network); Brigham and Women's Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IRB00249874
Record Dates: First submitted 2020-06-16; First posted 2020-06-17 (Actual); Results first posted 2021-11-09 (Actual); Last update posted 2021-11-09 (Actual); Status verified 2021-11

CONDITIONS: COVID-19
Keywords: coronavirus
MeSH Terms: conditions — COVID-19; Coronavirus Infections | interventions — crizanlizumab; Saline Solution

STUDY DESIGN:
Intervention Model Description: Double-blind, placebo-controlled, randomized interventional trial.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Crizanlizumab (Experimental): Crizanlizumab is a monoclonal antibody targeting P-selectin. Crizanlizumab 5.0 mg/kg in 100 ml IV once.
  Interventions: Drug: Crizanlizumab
- Placebo Saline (Active Comparator): 0.9% saline 100 ml IV once.
  Interventions: Other: 0.9% saline

INTERVENTIONS:
Drug: Crizanlizumab — Crizanlizumab 5.0 mg/kg in 100 ml IV once.
  Arms: Crizanlizumab
Other: 0.9% saline — 0.9% saline 100 ml IV once.
  Arms: Placebo Saline

SUMMARY:
The purpose of this trial is to test the efficacy and safety of crizanlizumab in patients hospitalized with COVID-19.

DETAILED DESCRIPTION:
Infection with severe acute respiratory syndrome (SARS) coronavirus 2 (CoV-2) causes coronavirus disease 2019 (COVID-19). The clinical course of COVID-19 is variable, and some patients develop severe pneumonia, multi-organ failure, and shock.

Severe COVID-19 is characterized by a hyper-inflammatory and hyper-thrombotic state. We propose that this state is caused by viral injury of the vascular endothelium, leading to endothelial release of von Willebrand Factor (VWF) and P-selectin, which in turn drive thrombosis and vascular inflammation.

Crizanlizumab is a monoclonal antibody that targets P-selectin. Crizanlizumab can decrease inflammation by binding to P-selectin, blocking leucocyte and platelet adherence to the vessel wall.

We now plan to test the safety and efficacy of crizanlizumab in decreasing biomarkers of inflammation and thrombosis in a placebo-controlled, double-blind randomized clinical trial

ELIGIBILITY:
Inclusion Criteria:

1. Willing to provide written informed consent
2. Willing to comply with all study procedures and be available for the duration of the study
3. Male or female ≥ 18 years of age
4. SARS-CoV-2 infection (COVID-19) within the past 10 d documented by laboratory test (nucleic acid test (NAT) or reverse transcriptase-polymerase chain reaction (RT-PCR))
5. Currently hospitalized
6. Symptoms of acute respiratory infection (at least one of the following: cough, fever > 37.5°C, dyspnea, sore throat, anosmia),
7. Radiographic evidence of pulmonary infiltrates
8. Requiring supplemental oxygen or the peripheral capillary oxygenation saturation (SpO2) < 94% on room air at screening
9. Elevated D-Dimer > 0.49 mg/L
10. Negative pregnancy test for females of childbearing potential

Exclusion Criteria:

1. Use of home oxygen at baseline
2. Current use of mechanical ventilation
3. Inability to provide consent
4. Do not intubate status
5. Prisoner or incarcerated
6. Pregnancy or Breast Feeding
7. Participation in other interventional therapy trials for COVID-19.
8. International normalized ratio (INR) > 3 or activated partial thromboplastin time (aPTT) > 60

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2020-07-09 (Actual); Primary Completion 2020-11-28 (Actual); Study Completion 2021-01-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Charles J Lowenstein, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Hospital, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ataga KI, Kutlar A, Kanter J, Liles D, Cancado R, Friedrisch J, Guthrie TH, Knight-Madden J, Alvarez OA, Gordeuk VR, Gualandro S, Colella MP, Smith WR, Rollins SA, Stocker JW, Rother RP. Crizanlizumab for the Prevention of Pain Crises in Sickle Cell Disease. N Engl J Med. 2017 Feb 2;376(5):429-439. doi: 10.1056/NEJMoa1611770. Epub 2016 Dec 3. PMID 27959701
- [Derived] Leucker TM, Osburn WO, Reventun P, Smith K, Claggett B, Kirwan BA, de Brouwer S, Williams MS, Gerstenblith G, Hager DN, Streiff MB, Solomon SD, Lowenstein CJ. Effect of Crizanlizumab, a P-Selectin Inhibitor, in COVID-19: A Placebo-Controlled, Randomized Trial. JACC Basic Transl Sci. 2021 Dec;6(12):935-945. doi: 10.1016/j.jacbts.2021.09.013. Epub 2021 Dec 8. PMID 34904132
- [Derived] Metkus TS, Sokoll LJ, Barth AS, Czarny MJ, Hays AG, Lowenstein CJ, Michos ED, Nolley EP, Post WS, Resar JR, Thiemann DR, Trost JC, Hasan RK. Myocardial Injury in Severe COVID-19 Compared With Non-COVID-19 Acute Respiratory Distress Syndrome. Circulation. 2021 Feb 9;143(6):553-565. doi: 10.1161/CIRCULATIONAHA.120.050543. Epub 2020 Nov 13. PMID 33186055

RESULTS

PARTICIPANT FLOW:
Recruitment Details: From July 15, 2020 through November 27, 2020, 583 patients were screened at 3 hospitals within the Johns Hopkins Health System. A total of 54 patients who fulfilled study entry criteria were randomized to receive crizanlizumab (n = 27) or placebo (n = 27).
Pre-assignment Details: Out of the 27 assigned to receive crizanlizumab, 2 did not receive crizanlizumab because of early discharge or early intubation. Out of the 27 assigned to receive placebo, 2 did not receive placebo because of early discharge or withdrawn consent.
Period: Overall Study
Arm/Group | Crizanlizumab | Placebo Saline
Started | 25 | 25
Completed | 22 | 20
Not Completed | 3 | 5
Not completed — follow-up blood draws missing | 3 | 5

BASELINE CHARACTERISTICS:
Population: Baseline characteristics data was collected for the 42 participants who completed the study.
Groups:
- Total: Total of all reporting groups
Arm/Group | Crizanlizumab | Placebo Saline | Total
Number analyzed (Participants) | 22 | 20 | 42
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 19 | 12 | 31
  >=65 years | 3 | 8 | 11
Age, Continuous [Mean (Standard Deviation); unit: years] | 58 (17.7) | 54.6 (13.4) | 56.2 (15.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 9 | 18
  Male | 13 | 11 | 24
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 14 | 6 | 20
  White | 8 | 13 | 21
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 22 | 20 | 42

OUTCOME MEASURES:

1. Primary Outcome: Soluble P-selectin Level
Description: Level of soluble P-selectin in ng/mL.
Time Frame: Day 3 after randomization or day of hospital discharge, whichever is earlier
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Crizanlizumab | Placebo Saline
Number analyzed (Participants) | 22 | 20
ng/mL | 7 (7) | 39 (18)

2. Secondary Outcome: Soluble P-selectin Level
Description: Level of soluble P-selectin in ng/mL.
Time Frame: Day 7 after randomization
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Crizanlizumab | Placebo Saline
Number analyzed (Participants) | 22 | 20
ng/mL | 10 (8) | 48 (17)

3. Secondary Outcome: Soluble P-selectin Level
Description: Level of soluble P-selectin in ng/mL.
Time Frame: Day 14 after randomization
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Crizanlizumab | Placebo Saline
Number analyzed (Participants) | 22 | 20
ng/mL | 12 (10) | 48 (24)

4. Secondary Outcome: D-dimer Level
Description: Level of D-dimer in mg/L.
Time Frame: Day 3 after randomization
Measure: Median (Inter-Quartile Range); unit: mg/L
Arm/Group | Crizanlizumab | Placebo Saline
Number analyzed (Participants) | 22 | 20
mg/L | 1.6 [0.7 to 2.8] | 0.7 [0.5 to 1.4]

5. Secondary Outcome: D-dimer Level
Description: Level of D-dimer in mg/L.
Time Frame: Day 7 after randomization
Measure: Median (Inter-Quartile Range); unit: mg/L
Arm/Group | Crizanlizumab | Placebo Saline
Number analyzed (Participants) | 22 | 20
mg/L | 1.6 [0.6 to 2.0] | 0.7 [0.5 to 0.8]

6. Secondary Outcome: D-dimer Level
Description: Level of D-dimer in mg/L.
Time Frame: Day 14 after randomization
Measure: Median (Inter-Quartile Range); unit: mg/L
Arm/Group | Crizanlizumab | Placebo Saline
Number analyzed (Participants) | 22 | 20
mg/L | 1.5 [0.5 to 1.9] | 0.7 [0.5 to 0.8]

7. Secondary Outcome: VWF Level
Description: Level of von Willebrand Factor (VWF) antigen in IU/mL.
Time Frame: Day 3 after randomization
Measure: Median (Inter-Quartile Range); unit: IU/mL
Arm/Group | Crizanlizumab | Placebo Saline
Number analyzed (Participants) | 22 | 20
IU/mL | 2.9 [1.9 to 4.9] | 2.8 [1.7 to 4.1]

8. Secondary Outcome: VWF Level
Description: Level of VWF antigen in IU/mL.
Time Frame: Day 7 after randomization
Measure: Median (Inter-Quartile Range); unit: IU/mL
Arm/Group | Crizanlizumab | Placebo Saline
Number analyzed (Participants) | 22 | 20
IU/mL | 3.9 [2.5 to 5.9] | 3.6 [2.1 to 6.8]

9. Secondary Outcome: VWF Level
Description: Level of VWF antigen in IU/mL.
Time Frame: Day 14 after randomization
Measure: Median (Inter-Quartile Range); unit: IU/mL
Arm/Group | Crizanlizumab | Placebo Saline
Number analyzed (Participants) | 22 | 20
IU/mL | 2.7 [1.9 to 4.2] | 4.6 [2.6 to 7.4]

10. Secondary Outcome: CRP Level
Description: Level of C-reactive protein (CRP) in mg/dL.
Time Frame: Day 3 after randomization
Measure: Median (Inter-Quartile Range); unit: mg/dL
Arm/Group | Crizanlizumab | Placebo Saline
Number analyzed (Participants) | 22 | 20
mg/dL | 4.4 [2.1 to 5.6] | 4.5 [1.2 to 6.9]

11. Secondary Outcome: CRP Level
Description: Level of C-reactive protein (CRP) in mg/dL.
Time Frame: Day 7 after randomization
Measure: Median (Inter-Quartile Range); unit: mg/dL
Arm/Group | Crizanlizumab | Placebo Saline
Number analyzed (Participants) | 22 | 20
mg/dL | 2.4 [1.1 to 4.9] | 2.1 [0.6 to 4.2]

12. Secondary Outcome: CRP Level
Description: Level of C-reactive protein (CRP) in mg/dL.
Time Frame: Day 14 after randomization
Measure: Median (Inter-Quartile Range); unit: mg/dL
Arm/Group | Crizanlizumab | Placebo Saline
Number analyzed (Participants) | 22 | 20
mg/dL | 2.5 [1.1 to 5.1] | 1.3 [0.6 to 4.9]

13. Secondary Outcome: Change in Clinical Status as Assessed by the World Health Organization (WHO) Ordinal Scale for Coronavirus Disease 2019 (COVID-19) Trials
Description: Change in the clinical status over 14 days as measured by an ordinal scale that is the first assessment of the clinical status on a given study day. The scale is as follows:
  0 = Uninfected; no viral RNA detected
  1. = Ambulatory; asymptomatic; viral RNA detected
  2. = Ambulatory; symptomatic; independent
  3. = Ambulatory; symptomatic; assistance needed
  4. = Hospitalized; no oxygen therapy
  5. = Hospitalized; oxygen by mask or nasal prongs
  6. = Hospitalized; oxygen by non-invasive ventilation (NIV) or high flow
  7. = Hospitalized; intubation and mechanical ventilation, partial pressure of oxygen / fraction of inspired oxygen (pO2/FIO2) ≥ 150 or oxygen saturation / FIO2 (SpO2/FIO2) ≥ 200
  8. = Hospitalized; intubation and mechanical ventilation, pO2/FIO2 < 150 or SpO2/FIO2 < 200 or vasopressors
  9. = Hospitalized; intubation and mechanical ventilation, pO2/FIO2 < 150 or SpO2/FIO2 < 200 and vasopressors, dialysis, or extracorporeal membrane oxygenation (ECMO)
  10. = Dead
Time Frame: Days 3, 7 and 14 after randomization
Measure: Count of Participants; unit: Participants
Arm/Group | Crizanlizumab | Placebo Saline
Number analyzed (Participants) | 22 | 20
Participants
  WHO Clinical Status: Day 3: </= 3 (discharged) | 3 | 2
  WHO Clinical Status: Day 3: 4 | 3 | 7
  WHO Clinical Status: Day 3: 5 | 13 | 7
  WHO Clinical Status: Day 3: 6 | 3 | 4
  WHO Clinical Status: Day 3: 7 | 0 | 0
  WHO Clinical Status: Day 3: 8 | 0 | 0
  WHO Clinical Status: Day 3: 9 | 0 | 0
  WHO Clinical Status: Day 3: 10 | 0 | 0
  WHO Clinical Status: Day 7: </= 3 (discharged) | 9 | 13
  WHO Clinical Status: Day 7: 4 | 5 | 3
  WHO Clinical Status: Day 7: 5 | 6 | 3
  WHO Clinical Status: Day 7: 6 | 1 | 1
  WHO Clinical Status: Day 7: 7 | 1 | 0
  WHO Clinical Status: Day 7: 8 | 0 | 0
  WHO Clinical Status: Day 7: 9 | 0 | 0
  WHO Clinical Status: Day 7: 10 | 0 | 0
  WHO Clinical Status: Day 14: </= 3 (discharged) | 21 | 19
  WHO Clinical Status: Day 14: 4 | 0 | 0
  WHO Clinical Status: Day 14: 5 | 0 | 0
  WHO Clinical Status: Day 14: 6 | 1 | 0
  WHO Clinical Status: Day 14: 7 | 0 | 0
  WHO Clinical Status: Day 14: 8 | 0 | 1
  WHO Clinical Status: Day 14: 9 | 0 | 0
  WHO Clinical Status: Day 14: 10 | 0 | 0

14. Secondary Outcome: Time to Hospital Discharge
Description: Time (days) to hospital discharge
Time Frame: Up to 30 days after randomization
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Crizanlizumab | Placebo Saline
Number analyzed (Participants) | 22 | 20
days | 8.1 (4.4) | 6.2 (3.2)

15. Secondary Outcome: Safety of Crizanlizumab as Assessed by Adverse Events
Description: Safety of crizanlizumab will by assessed by adverse events, serious adverse events, and suspected unexpected serious adverse reactions.
Time Frame: Up to day 14 after randomization
Measure: Number; unit: total adverse events
Arm/Group | Crizanlizumab | Placebo Saline
Number analyzed (Participants) | 25 | 25
total adverse events | 7 | 6

ADVERSE EVENTS:
Time Frame: 30 days
Arm/Group | Crizanlizumab | Placebo Saline
All-Cause Mortality (participants affected / at risk) | 0/25 | 0/25
Serious Adverse Events (participants affected / at risk) | 0/25 | 1/25
Other Adverse Events (participants affected / at risk) | 7/25 | 5/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Crizanlizumab (N=25) | Placebo Saline (N=25)
multi-organ failure (General disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Crizanlizumab (N=25) | Placebo Saline (N=25)
Headache (Nervous system disorders) | 1 (1) | 0 (0)
Venous thrombembolism (Vascular disorders) | 1 (1) | 1 (1)
Altered mental status (Nervous system disorders) | 1 (1) | 0 (0)
Chest pain (Cardiac disorders) | 2 (2) | 1 (1)
Urinary tract infection (Renal and urinary disorders) | 0 (0) | 1 (1)
Diarrhea (Metabolism and nutrition disorders) | 1 (1) | 2 (2)
Dark and Infrequent Urination (Renal and urinary disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-12-14): https://cdn.clinicaltrials.gov/large-docs/84/NCT04435184/Prot_SAP_000.pdf